CLINICAL TRIAL: NCT03495531
Title: Virtual Reality Obstetrics Phase 1 & Phase 2 Prospective Study
Brief Title: Virtual Reality in Obstetric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 45042
Record Dates: First submitted 2018-03-15; First posted 2018-04-12 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2020-08

CONDITIONS: Obstetric Pain; Pain
Keywords: virtual reality; obstetrics; labor procedures; regional anesthesia
MeSH Terms: conditions — Labor Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care
- VR Use (Experimental): Obstetrics patients who use virtual reality
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality headset with calming scenery
  Arms: VR Use

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality headset) are more effective than the standard of care (i.e., no technology based distraction) for preventing anxiety and pain scores in women who are undergoing child laboring procedures. The anticipated primary outcome will be a reduction of pregnant females overall anxiety and pain scores before and after such procedure(s), including but not limited to epidural/combined spinal epidural (CSE), IV placement and/or labor.

DETAILED DESCRIPTION:
Phase 1 There will be 3 stages that are sequentially and chronologically timed in order to asses the efficacy of Virtual Reality (VR) in the reducing epidural/combined spinal-epidural (CSE) related pain and anxiety at every stage. Phase 1 is the development phase where the focus is primarily on feasibility for Phase 2. The exclusion criteria will remain the same for all the stages and includes (i) participants and patients who do not consent (ii) have significant cognitive impairment (iii) have a history of severe motion sickness (iv) currently have nausea (v) currently experiencing seizures (vi) have visual problems(vii) are clinically unstable or require urgent/emergent intervention and/or (viii) are Non-English Speaking. Inclusion criteria is that females are (i)18 years or older and (ii) who had either have a history of, planning to have, or currently having an child laboring related procedures such as IV placement, epidural/CSE placement and/or labor.

(Stage 1) The first stage will include 10 females who are not pregnant, but have previously have at least undergone one labor epidural/CSE in the past. These mothers will be approached by a clinician or healthcare provider at Lucille Packard Children's Hospital (LPCH) outpatient surgical procedures as they wait for their child. If they are interested, the healthcare provider will let the research staff know of the eligible participant. During the mother's wait time, the research assistant will review the study, go over the consent forms and answer any questions in regards to their participation in the study. Once the participant is consented into the study, the research assistant will provide the participant with a survey regarding their recall pain and anxiety (refer to section 16) during their most recent epidural (if participant has had previously had more than one). The research assistant will then provide the participant with a VR headset and guide them through a series of VR scenery, shortly after the VR simulation the participant will be given a feedback survey in regards to their VR experience.

(Stage 2) The second stage will include 10 different females who are currently either in their second or third trimester of pregnancy. These mothers will be approached by a clinician or healthcare provider during their visits to obstetrics clinic at LPCH and Stanford Health Care (SHC) facilities. If they are interested, the healthcare provider will let the research staff know of the eligible participant. During the patients wait time, the research assistant will review the study, go over the consent forms and answer any questions in regards to their participation in the study. Once the participant is consented into the study, the research assistant will provide the participant with a survey regarding their current anxiety about labor and epidural/CSE placement. The research assistant will then provide the participant with a VR headset and guide them through a series of VR scenery, shortly after the VR simulation the participant will be given a feedback survey in regards to their VR experience. Since this cohort can give the investigators better guidance of intolerance (i.e nausea and dizziness) during VR simulation, the clinicians and research providers have come up with a safety threshold: if more than 20 percent of patients answer to a score of 4 or higher on questions regarding nausea and dizziness, the clinicians and health care providers will have to go back and iterate on VR software and repeat the previous stage before moving on stage 3.

(Stage 3) If stage 2 outcomes meet the investigator's criteria, the clinical team will move on to the last stage of 10 different females who are currently in labor and planning on undergoing an epidural for child-laboring. These mothers will be approached by their obstetric anesthesiologist during their first anesthesia consult after being admitted into LPCH labor and delivery facilities. If they are interested, the anesthesiologist will let the research staff know of the eligible participant. During the patients wait time, the research assistant and/or anesthesiologist will review the study, go over the consent forms and answer any questions in regards to their participation in the study. Once the patient is consented into the study, the research assistant and/or anesthesiologist will provide the participant with a survey regarding their pre-epidural anxiety and pain scores. The anesthesiologist and/or research assistant will then provide the laboring mother with a VR headset during epidural/CSE placement by anesthesiologist. Depending on the mother's laboring timeline, if possible, mother will receive VR feedback survey and post-epidural anxiety and pain scores. If not, mothers will receive post-epidural anxiety and pain scores where they recall these scores and fill out VR feedback survey postpartum.

Phase 2:

Based on preliminary and feasibility data from Phase 1, if the clinicians and study personnel find it appropriate, the study will move on to Phase 2, a randomized prospective clinical trial focused more broadly on technology based distractions (VR headsets) in comparison to standard of care (no VR use) in obstetric patients for preventing anxiety and pain during various laboring procedures. These laboring procedures include but are not limited to IV, epidural/CSE placement and/or child-labor. Inclusion and exclusion criteria will remain the same as Phase 1. For Phase 2, the study personnel expect to enroll 200 mothers who've been admitted into LPCH labor and delivery services. These mothers will be approached by their obstetric anesthesiologist during their first anesthesia consult after being admitted into LPCH labor and delivery facilities. If they are interested, the anesthesiologist will let the research staff know of the eligible participant. During the patients wait time, the research assistant and/or anesthesiologist will review the study, go over the consent forms and answer any questions in regards to their participation in the study. Once the patient is consented into the study, the research assistant and/or anesthesiologist will provide the participant with a survey regarding their pre-procedure anxiety and pain scores. Depending on a randomized generator, mothers will either be placed into VR use group during procedure or standard of care (no VR use). If mother falls under VR group, the anesthesiologist and/or research assistant will then provide the laboring mother with a VR headset during procedure by anesthesiologist. Depending on the mother's laboring timeline, if possible, mother will receive VR feedback survey and post- procedure anxiety and pain scores. If not, mothers will receive post-epidural anxiety and pain scores where they recall these scores and fill out VR feedback survey postpartum. If mother falls under control group, mother will undergo standard of care and receive pre and post- pain and anxiety surveys regarding procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Able to consent
* Obstetric patients who had either have a history of, planning to have, or currently having an child laboring related procedures such as IV placement, epidural/CSE placement and/or labor.

Exclusion Criteria:

* Inclusion Criteria:
* Age 18 and over
* Able to consent
* Obstetric patients who had either have a history of, planning to have, or currently having an child laboring related procedures such as IV placement, epidural/CSE placement and/or labor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Obstetrics patients undergoing various child-laboring procedures
Enrollment: 60 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Virtual Reality vs Standard Of Care | Throughout Study Completion, an average of 1-2 years.
  Investigators hope to determine if technology based distractions (VR headsets) are more effective than standard of care in obstetric patients for preventing high anxiety and pain during laboring procedures. This will be assessed using pre-/post- surveys.

SECONDARY OUTCOMES:
Parent/Patient Assessment of Virtual Reality Software | Evaluated post procedure, between 5-60 minutes after such procedure.
  As a secondary aim of the study, the investigators seek to determine if the use of technology based distraction (i.e virtual reality) will result in higher patient satisfaction as well as evaluating which techniques or software scenery are the most effective for relaxation.
Epidural/Combined Spinal-Epidural Dosing Requirements | Duration of procedure, which is generally less than 2 hours
  Assessment of cumulative epidural dosing and the duration of epidural analgesia of participants through child-laboring procedures.
Overall Change in Pain Scores Using Virtual Reality | Duration of procedure, which is generally less than 2 hours
  Comparing whether passive or active interventions using VR are more effective in decreasing overall pain scores in participants by comparing pre-/post- procedure survey answers.
Overall Change in Anxiety Scores Using Virtual Reality | Duration of procedure, which is generally less than 2 hours
  Comparing whether passive or active interventions using VR are more effective in decreasing overall anxiety scores in participants by comparing pre-/post- procedure survey answers.

CONTACTS AND LOCATIONS:
Locations (1):
- LPCH/SHC, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified and used collectively for research analysis.

REFERENCES:
- [Result] Poggi L, Goutaudier N, Sejourne N, Chabrol H. When Fear of Childbirth is Pathological: The Fear Continuum. Matern Child Health J. 2018 May;22(5):772-778. doi: 10.1007/s10995-018-2447-8. PMID 29484511
- [Result] Demsar K, Svetina M, Verdenik I, Tul N, Blickstein I, Globevnik Velikonja V. Tokophobia (fear of childbirth): prevalence and risk factors. J Perinat Med. 2018 Feb 23;46(2):151-154. doi: 10.1515/jpm-2016-0282. PMID 28379837
- [Result] Wulff V, Hepp P, Fehm T, Schaal NK. Music in Obstetrics: An Intervention Option to Reduce Tension, Pain and Stress. Geburtshilfe Frauenheilkd. 2017 Sep;77(9):967-975. doi: 10.1055/s-0043-118414. Epub 2017 Sep 25. PMID 28959060
- [Result] Gokyildiz Surucu S, Ozturk M, Avcibay Vurgec B, Alan S, Akbas M. The effect of music on pain and anxiety of women during labour on first time pregnancy: A study from Turkey. Complement Ther Clin Pract. 2018 Feb;30:96-102. doi: 10.1016/j.ctcp.2017.12.015. Epub 2017 Dec 19. PMID 29389487
- [Result] Anderson AP, Mayer MD, Fellows AM, Cowan DR, Hegel MT, Buckey JC. Relaxation with Immersive Natural Scenes Presented Using Virtual Reality. Aerosp Med Hum Perform. 2017 Jun 1;88(6):520-526. doi: 10.3357/AMHP.4747.2017. PMID 28539139
- [Result] Hoffman HG, Seibel EJ, Richards TL, Furness TA, Patterson DR, Sharar SR. Virtual reality helmet display quality influences the magnitude of virtual reality analgesia. J Pain. 2006 Nov;7(11):843-50. doi: 10.1016/j.jpain.2006.04.006. PMID 17074626
- [Result] Dahlquist LM, Weiss KE, Law EF, Sil S, Herbert LJ, Horn SB, Wohlheiter K, Ackerman CS. Effects of videogame distraction and a virtual reality type head-mounted display helmet on cold pressor pain in young elementary school-aged children. J Pediatr Psychol. 2010 Jul;35(6):617-25. doi: 10.1093/jpepsy/jsp082. Epub 2009 Sep 28. PMID 19786489